CLINICAL TRIAL: NCT07305415
Title: Integrative Therapeutic Programme to Regulate Expressed Emotions Among Informal Caregivers of People With Dementia: a Pilot Randomized Controlled Trial
Brief Title: Integrative Therapeutic Programme to Regulate Expressed Emotions Among Informal Caregivers of People With Dementia
Acronym: COPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Proferssor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COPE
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: BPSD (Behavioral and Psycological Symptoms of Dementia); Expressed Emotion; Depressive Symptom; Caregiving Stress
Keywords: BPSD; behavioral and psychological symptoms of dementia; Expressed Emotion; Dementia caregivers; Dementia caregiving; preceived stress; caregiver depression; caregiving stress; caregiving relationship; dyadic care relationship
MeSH Terms: conditions — Behavior; Depression; Caregiver Burden | interventions — Mindfulness; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPE Intervention Group (Experimental): COPE is a 6-week group-based programme comprising one face-to-face workshop (4 caregivers per group) and five online sessions (4 caregivers per group) delivered via Zoom. The COPE programme integrates the strategies from cognitive behavioral therapy (CBT), emotional-focused mindfulness therapy and social skill training to improve the expressed emotion (EE) of the caregivers, with the focus to ameliorate negative causal attrition of BPSD, increase emotional regulation and enhance social interaction skills with PwD. The group size of 4 is used to optimize the social interactions between the peer caregivers. The first session will adopt a face-to-face mode to better develop their rapport with each other, and to facilitate their self-reflection and disclosure on their social interaction with the care recipients in day-to-day caregiving.
  Interventions: Behavioral: Caregivers Of dementia Processing Emotions (COPE)
- Control group (No Intervention): Participants in the waitlist control group, in comparison to those in the intervention group who receive treatment immediately, are placed on a waiting list and receive the same set of intervention sessions after the formal trial. This approach ensures participants have equal opportunity to receive treatment while strengthening the study's validity and overall quality by maximally controlling for potential confounding variables and biases.

INTERVENTIONS:
Behavioral: Caregivers Of dementia Processing Emotions (COPE) — This is the first study to develop an easily accessible and feasible intervention programme, namely the Caregivers Of dementia Processing Emotions (COPE), to primarily reduce expressed emotion (EE) in family caregivers of PwD via processing one's attributional biases, dysregulated emotion, dysfunctional social dynamics using an integrative therapy. By displacing these negative thoughts and emotions, the integrative therapy has great potential to reduce the depressive symptoms in caregivers and thus mitigate their perceived stress from BPSD. In addition, the interactive social dynamics in the dementia caregiving context can be improved.
  Other Names: COPE; Mindfulness and Cognitive Behavioral Therapy
  Arms: COPE Intervention Group

SUMMARY:
The dual-modal (face-to-face and online approaches), client-customized Caregivers Of dementia Processing Emotions (COPE) programme aims to

1. reduce caregivers' Expressed Emotion (EE),
2. reduce caregivers' depressive symptoms,
3. reduce the behaviourally interactive social dynamic of maladaptation (i.e., dysfunctional dyadic relationship and quality of care), and
4. improve caregivers' perceived stress from PwD's Behavioral and Psychological Symptoms of Dementia (BPSD).

Researchers will compare COPE to a control group (standard therapy) to examine how effective the COPE programme is.

Participants will take part in:

Pretest prior to COPE implementation Post-test after COPE completion Follow up test in 3 months after COPE completion

DETAILED DESCRIPTION:
Primary Purpose Prevention: Assessing the effectiveness of a novel intervention for preventing the development of negative outcomes in caregivers as a result of managing behavioral psychological symptoms of dementia.

Interventional Study Model:

Parallel: Participants are assigned to one of two groups in parallel for the duration of the study.

Model Description:

Participants are assigned to either COPE group or control group on a random basis. Baseline data are collected either face-to-face or online before the implementation. After six weeks of implementation, post-test data will be collected either face-to-face or online. Three months after post-test, follow-up data will be collected either face-to-face or online.

Number of Arms:

Two total arms, one for the COPE intervention group and one for the standard therapy control group.

Masking:

Participants Outcomes Assessors

Allocation:

Randomized: Participants are assigned to intervention groups by chance

Enrollment:

At least 56 subjects are needed for the two arms to allow the most accurate variance estimation for intervention of small to medium standardised effect size (0.2-0.6) at 80% power and 5% level of significance, with a 10% attrition rate. The social workers in the Psychogeriatric Day Hospital (Queen Mary Hospital) will refer the potential family caregivers of PwD to the RA for eligibility screening. Informed consent will be obtained accordingly.

ELIGIBILITY:
Inclusion Criteria:

* (1) With a high level of EE as indicated by a cut-off score of 35 or above on the Family Attitude Scale (Chinese version; FAS-C)
* (2) Provides care at least 4 hours per day
* (3) Consent to participate
* (4) No acute psychiatric illness

Exclusion Criteria:

* (1) With a score below 35 on the Family Attitude Scale (Chinese version; FAS-C)
* (2) Provides care no more than 4 hours per day
* (3) Does not consent to participate
* (4) With acute psychiatric illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Family Attitude Scale- Chinese Version | From enrollment to the end of intervention at 7 weeks and end of study at 20 weeks.
  Measure caregivers' expressed emotions (EE) (i.e., criticism and hostility) held towards the PwD.

SECONDARY OUTCOMES:
Center of Epidemiological Studies of Depression Revised - Chinese Version | From enrollment to the end of intervention at 7 weeks and end of study at 20 weeks.
  Assess caregivers' depression
Dyadic Relationship Scale - Chinese Version | From enrollment to the end of intervention at 7 weeks and end of study at 20 weeks.
  Evaluate caregivers' perspective of dyadic and family relationships in their daily caregiving activities
Interaction Quality Scale - Chinese Version | From enrollment to the end of intervention at 7 weeks and end of study at 20 weeks.
  Measure the quality of care.
Neuropsychiatric Inventory - Chinese Version | From enrollment to the end of intervention at 7 weeks and end of study at 20 weeks.
  Assess the severity of BPSD manifested in PwD reported by their caregivers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen S, Lin K, Wang H, Yamakawa M, Makimoto K, Liao X. Reliability and structural validity of the Chinese version of the Neuropsychiatric Inventory, Nursing Home version. Psychogeriatrics. 2018 Mar;18(2):113-122. doi: 10.1111/psyg.12292. Epub 2018 Feb 6. PMID 29409164
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Joseph NT, Kamarck TW, Muldoon MF, Manuck SB. Daily marital interaction quality and carotid artery intima-medial thickness in healthy middle-aged adults. Psychosom Med. 2014 Jun;76(5):347-54. doi: 10.1097/PSY.0000000000000071. PMID 24915293
- [Background] Cundiff JM, Kamarck TW, Manuck SB. Daily Interpersonal Experience Partially Explains the Association Between Social Rank and Physical Health. Ann Behav Med. 2016 Dec;50(6):854-861. doi: 10.1007/s12160-016-9811-y. PMID 27333896
- [Background] Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID 18192628
- [Background] Zhang Y, Ting RZ, Lam MH, Lam SP, Yeung RO, Nan H, Ozaki R, Luk AO, Kong AP, Wing YK, Sartorius N, Chan JC. Measuring depression with CES-D in Chinese patients with type 2 diabetes: the validity and its comparison to PHQ-9. BMC Psychiatry. 2015 Aug 18;15:198. doi: 10.1186/s12888-015-0580-0. PMID 26281832
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement. 1977;1(3):385-401.
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Moon H, Adams KB. The effectiveness of dyadic interventions for people with dementia and their caregivers. Dementia (London). 2013 Nov;12(6):821-39. doi: 10.1177/1471301212447026. Epub 2012 May 21. PMID 24337642
- [Background] Van Humbeeck G, Van Audenhove Ch, De Hert M, Pieters G, Storms G. Expressed emotion: a review of assessment instruments. Clin Psychol Rev. 2002 Apr;22(3):323-43. doi: 10.1016/s0272-7358(01)00098-8. PMID 17201189
- [Background] Kavanagh DJ, O'Halloran P, Manicavasagar V, Clark D, Piatkowska O, Tennant C, Rosen A. The Family Attitude Scale: reliability and validity of a new scale for measuring the emotional climate of families. Psychiatry Res. 1997 May 30;70(3):185-95. doi: 10.1016/s0165-1781(97)00033-4. PMID 9211580
- [Background] Rothbaum BO, Meadows EA, Resick P, Foy DW. Cognitive-behavioral therapy. Published online 2000.
- [Background] Bejan A, Merkx GW. Constructal Theory of Social Dynamics. Springer London NetLibrary, Inc. [distributor]
- [Background] Steffen AM, Gant JR. A telehealth behavioral coaching intervention for neurocognitive disorder family carers. Int J Geriatr Psychiatry. 2016 Feb;31(2):195-203. doi: 10.1002/gps.4312. Epub 2015 Jun 15. PMID 26077904
- [Background] Moore RC, Chattillion EA, Ceglowski J, Ho J, von Kanel R, Mills PJ, Ziegler MG, Patterson TL, Grant I, Mausbach BT. A randomized clinical trial of Behavioral Activation (BA) therapy for improving psychological and physical health in dementia caregivers: results of the Pleasant Events Program (PEP). Behav Res Ther. 2013 Oct;51(10):623-32. doi: 10.1016/j.brat.2013.07.005. Epub 2013 Jul 19. PMID 23916631
- [Background] Bjorge H, Kvaal K, Ulstein I. The effect of psychosocial support on caregivers' perceived criticism and emotional over-involvement of persons with dementia: an assessor-blinded randomized controlled trial. BMC Health Serv Res. 2019 Oct 24;19(1):744. doi: 10.1186/s12913-019-4551-x. PMID 31651321
- [Background] Wiegelmann H, Speller S, Verhaert LM, Schirra-Weirich L, Wolf-Ostermann K. Psychosocial interventions to support the mental health of informal caregivers of persons living with dementia - a systematic literature review. BMC Geriatr. 2021 Feb 1;21(1):94. doi: 10.1186/s12877-021-02020-4. PMID 33526012
- [Background] Scott JL, Dawkins S, Quinn MG, Sanderson K, Elliott KE, Stirling C, Schuz B, Robinson A. Caring for the carer: a systematic review of pure technology-based cognitive behavioral therapy (TB-CBT) interventions for dementia carers. Aging Ment Health. 2016 Aug;20(8):793-803. doi: 10.1080/13607863.2015.1040724. Epub 2015 May 15. PMID 25978672
- [Background] Kovach CR, Noonan PE, Schlidt AM, Wells T. A model of consequences of need-driven, dementia-compromised behavior. J Nurs Scholarsh. 2005;37(2):134-40; discussion 140. doi: 10.1111/j.1547-5069.2005.00025_1.x. PMID 15960057
- [Background] Tarrier N, Barrowclough C, Ward J, Donaldson C, Burns A, Gregg L. Expressed emotion and attributions in the carers of patients with Alzheimer's disease: the effect on carer burden. J Abnorm Psychol. 2002 May;111(2):340-9. doi: 10.1037//0021-843x.111.2.340. PMID 12003455
- [Background] Hooley JM, Richters JE. Expressed emotion: A developmental perspective. In: Emotion, Cognition, and Representation. Rochester symposium on developmental psychopathology, Vol. 6. University of Rochester Press; 1995:133-166.
- [Background] Kelly RB, Zyzanski SJ, Alemagno SA. Prediction of motivation and behavior change following health promotion: role of health beliefs, social support, and self-efficacy. Soc Sci Med. 1991;32(3):311-20. doi: 10.1016/0277-9536(91)90109-p. PMID 2024141
- [Background] Weiner B. An Attributional Theory of Motivation and Emotion. Springer Science & Business Media; 2012.
- [Background] Weiner B. A cognitive (attribution)-emotion-action model of motivated behavior: An analysis of judgments of help-giving. Journal of Personality and Social psychology. 1980;39(2):186.
- [Background] Zhang S, Ying X, Fang S, Wang W, Zhu X, Dong Y, He M, Chang A, Sun J. The influence path of caregivers' positive aspects, expressed emotion and coping style on behavioral and psychological symptoms of dementia. Geriatr Nurs. 2022 Mar-Apr;44:143-150. doi: 10.1016/j.gerinurse.2022.01.013. Epub 2022 Feb 12. PMID 35158171
- [Background] Yu DS, Kwok T, Choy J, Kavanagh DJ. Measuring the expressed emotion in Chinese family caregivers of persons with dementia: Validation of a Chinese version of the Family Attitude Scale. Int J Nurs Stud. 2016 Mar;55:50-9. doi: 10.1016/j.ijnurstu.2015.11.005. Epub 2015 Dec 17. PMID 26742605
- [Background] Li CY, Lewis FM. Expressed emotion and depression in caregivers of older adults with dementia: results from Taiwan. Aging Ment Health. 2013;17(8):924-9. doi: 10.1080/13607863.2013.814098. Epub 2013 Jul 4. PMID 23826863
- [Background] Safavi R, Berry K, Wearden A. Expressed Emotion in relatives of persons with dementia: a systematic review and meta-analysis. Aging Ment Health. 2017 Feb;21(2):113-124. doi: 10.1080/13607863.2015.1111863. Epub 2015 Nov 16. PMID 26569025
- [Background] Li CY, Murray M. A review of conceptualisation of expressed emotion in caregivers of older adults with dementia. J Clin Nurs. 2015 Feb;24(3-4):332-43. doi: 10.1111/jocn.12619. Epub 2014 May 9. PMID 24811189
- [Background] Friedman EM, Kennedy DP. Typologies of Dementia Caregiver Support Networks: A Pilot Study. Gerontologist. 2021 Nov 15;61(8):1221-1230. doi: 10.1093/geront/gnab013. PMID 33585929
- [Background] National Alliance for Caregiving and the Alzheimer's Association. Dementia Caregiving in the U.S. National Alliance for Caregiving and the Alzheimer's Association; 2017. https://www.caregiving.org/wp-content/uploads/2020/05/Dementia-Caregiving-Report 2017_Research-Recommendations_FINAL.pdf
- [Background] Alzheimer's Association. 2018 Alzheimer's disease facts and figures. Alzheimer's & Dementia. 2018;14(3):367-429.
- [Background] Kales HC, Gitlin LN, Lyketsos CG. Assessment and management of behavioral and psychological symptoms of dementia. BMJ. 2015 Mar 2;350:h369. doi: 10.1136/bmj.h369. PMID 25731881
- [Background] Scassellati C, Ciani M, Maj C, Geroldi C, Zanetti O, Gennarelli M, Bonvicini C. Behavioral and Psychological Symptoms of Dementia (BPSD): Clinical Characterization and Genetic Correlates in an Italian Alzheimer's Disease Cohort. J Pers Med. 2020 Aug 14;10(3):90. doi: 10.3390/jpm10030090. PMID 32823921
- [Background] Cao Q, Tan CC, Xu W, Hu H, Cao XP, Dong Q, Tan L, Yu JT. The Prevalence of Dementia: A Systematic Review and Meta-Analysis. J Alzheimers Dis. 2020;73(3):1157-1166. doi: 10.3233/JAD-191092. PMID 31884487
- [Background] Alzheimer's Association. 2022 Alzheimer's Disease Facts and Figures. More Than Normal Aging: Understanding Mild Cognitive Impairment. Published online 2022.